CLINICAL TRIAL: NCT05191875
Title: Gastrointestinal Preparation and Efficacy of Saccharomyces Boulardii as a Pre-treatment for Helicobacter Pylori Rescue Therapy
Brief Title: Saccharomyces Boulardii as Pretreatment Before Rescue Therapy of Helicobacter Pylori
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: xucanxia
Record Dates: First submitted 2021-12-26; First posted 2022-01-14 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-01

CONDITIONS: Helicobacter Pylori Infection
Keywords: Saccharomyces boulardii Helicobacter pylori rescue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 of stage I (Experimental): 14-day therapy：Saccharomyces boulardii. 500mg b.i.d
  Interventions: Drug: Saccharomyces Boulardii 250 MG
- group 2 of stage I (No Intervention): Observe for one month before treatment
- stage 2 (Other): 14-day therapy：Ilaprazole. 5mg b.i.d Doxycycline. 0.1g b.i.d Furazolidone. 0.1g b.i.d Colloidal Bismuth Tartrate . 220mg b.i.d
  Interventions: Drug: Ilaprazole.Doxycycline. Furazolidone. Colloidal Bismuth Tartrate

INTERVENTIONS:
Drug: Saccharomyces Boulardii 250 MG — Saccharomyces Boulardii:
  0.25 g * 6, Produced by The French encyclopedia pharmaceutical Factory
  Other Names: treatment drugs of stage I
  Arms: group 1 of stage I
Drug: Ilaprazole.Doxycycline. Furazolidone. Colloidal Bismuth Tartrate — Ilaprazole:
  5mg*6, produced by Livzon Pharmaceutical Group Inc
  Doxycycline:
  0.1 g * 10, produced by Jiangsu Yongxin Ltd.
  Furazolidone:
  0.1g*100 produced by Tianjin Lisheng Pharmaceutical Co., LTD
  Colloidal Bismuth Tartrate:
  55 mg * 36,produced by Shanxi Xinbaoyuan Pharmaceutical Co., LTD
  Other Names: treatment drugs of stage II
  Arms: stage 2

SUMMARY:
The increasing rate of drug resistance in often leads to eradication failure and the need for rescue therapy, and it is of great significance to explore new rescue therapeutic regimens. In this study, we observed the efficacy of rescue treatment of Helicobacter pylori (H.pylori) with Saccharomyces boulardii (S.boulardii) alone. the primary outcome of the trial was the eradication rate, and the secondary outcome was the incidence of adverse events.

DETAILED DESCRIPTION:
Background: Helicobacter pylori(H.pylori)infection is a common bacterial infection that causes chronic gastritis, peptic ulcer, MALT lymphoma, gastric cancer, and other gastrointestinal diseases. and has been classified as a group 1 biologic carcinogen with a prevalence of about 50% population in china. In recent years, with the massive use of antibiotics, poor patient compliance, and irregular drug use, the side effects associated with drugs have increased and have led to the development of antibiotic-resistant bacteria and a gradual increase in refractory H.pylori infections, researchers have been searching for a safe, effective and simple treatment for H. pylori.

Methods: The patient come from the department of Gastroenterology, Xiangya Third Hospital, Central South University. After obtaining informed consent, patients is randomly divided into a study group and a control group. The study group (n=100) is divided into two stages of treatment, starting with Saccharomyces boulardii monnotherapy for 14 days, Patients who are still positive on reexamination after 4 weeks of stopping the drug continue with bismuth quadruple therapy. As for the control group (n=100), patients is observed for 4 weeks without any gastric drugs as well as antibiotics, and those who were still positive on retest after 4 weeks continued with bismuth quadruple therapy. We observe the eradication rate of patients and the occurrence of adverse effects during the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 to 65 years, of either sex
2. patients with a diagnosis of Hp infection
3. patients who have failed treatment for Hp infection
4. not taking acid-suppressing medications (PPI or H2 blockers) within the last 2 weeks
5. who have not used antibiotics and/or bismuth within the last 4 weeks
6. understand and are willing to participate in this clinical trial and provide a signed informed consent form.

Exclusion Criteria:

1. those with a history of drug allergy
2. those with severe cardiac, hepatic, pulmonary, and renal insufficiencies
3. those with a recent history of gastrointestinal hemorrhage, obstruction, perforation, tumors, and other serious organic diseases of the gastrointestinal tract
4. those with mental illness, psychological disorders that cannot be expressed normally
5. those who are pregnant, lactating, or planning to have children in the near future during the study period.
6. those who are not suitable for clinical trials and those who cannot cooperate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-23 (Actual)

PRIMARY OUTCOMES:
The eradication rate of H. pylori infection | Visit period 2 (day 42±3)
  Evaluated by 13C-urea breath test (13C-UBT), or 14C-urea breath test (14C-UBT).

SECONDARY OUTCOMES:
Adverse events | Visit period 1 (day 14±1), Visit period 2 (day 28±1)
  Follow-up of patients' adverse reactions by telephone and at the gastroenterology clinic

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No